CLINICAL TRIAL: NCT03002818
Title: Quality of Life Measurement Using Wrist Actigraphy in HCV Genotype 1 Infected, Treatment naïve Patients Suffering From Fatigue and Receiving Ombitasvir, Paritaprevir, and Ritonavir Tablets and Dasabuvir Tablets (Viekirax®/Exviera®; 3D Regimen): The HEMATITE Study
Brief Title: Quality of Life Measurement in Treatment Naïve Patients With Hepatitis C Virus (HCV) Genotype 1 (GT1) Suffering From Fatigue and Receiving Ombitasvir, Paritaprevir, and Ritonavir and Dasabuvir (Viekirax®/Exviera®)
Acronym: HEMATITE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-272
Record Dates: First submitted 2016-12-15; First posted 2016-12-26 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2018-05

CONDITIONS: Chronic Hepatitis C Virus (HCV)
Keywords: Chronic Hepatitis C (HCV); Genotype 1; Paritaprevir; Ritonavir; ombitasvir; Dasabuvir; Sustained Virological Response
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HCV Genotype 1 Participants: Participants receiving paritaprevir/ritonavir/ombitasvir with dasabuvir (Viekirax®/Exviera®, 3D regimen)

SUMMARY:
This is an observational, prospective, open-label, single-arm, multicenter, real-life study designed to observe the impact of paritaprevir/ritonavir/ombitasvir with dasabuvir regimen (Viekirax®/Exviera®, 3D regimen) on total daytime physical activity and fatigue in participants with HCV GT1.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve participants
* Mono-infected participants with chronic HCV GT1
* Non-cirrhotic participants
* Participants with debilitating fatigue (Fatigue Severity Scale [FSS] greater than or equal to 4)

Exclusion Criteria:

* Participants with sources of fatigue other than HCV (especially, severe depression, cancer and hormonal disorders causing clinically significant fatigue)
* Participants with conditions that do not allow to adhere to protocol and use of the device at investigator's discretion
* Participants who are wheelchair dependent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CHC, genotype 1, receiving paritaprevir/ritonavir/ombitasvir with dasabuvir regimen (3D regimen)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (5):
- Switzerland (5):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital, Universitaetsklin, Bern
  - Fondazione Epatocentro Ticino, Lugano
  - Hopital Neuchatelois, Neuchâtel
  - Universitaetsspital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Semmo N, Mullhaupt B, Ruckstuhl L, Magenta L, Clerc O, Torgler R, Semela D. A prospective, multicenter, post-marketing observational study to measure the quality of life of HCV genotype 1 infected, treatment naive patients suffering from fatigue and receiving 3D regimen: The HEMATITE study. PLoS One. 2020 Nov 4;15(11):e0241267. doi: 10.1371/journal.pone.0241267. eCollection 2020. PMID 33147283
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Hepatitis C Virus (HCV) Genotype 1 Participants: Participants receiving paritaprevir/ritonavir/ombitasvir with dasabuvir (Viekirax®/Exviera®, 3D regimen)
Period: Overall Study
Arm/Group | Hepatitis C Virus (HCV) Genotype 1 Participants
Started (eligible participants who received 3D regimen at least once) | 41
Completed | 40
Not Completed | 1
Not completed — Decision of the investigator | 1

BASELINE CHARACTERISTICS:
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 41
Mean Daytime Physical Activity [Mean (Standard Deviation); unit: day-counts] — Mean daytime physical activity for 2 eligible weeks (10 working days) prior to the assessment day was derived from a wrist-worn activity tracker (ActiGraph GT9X Link), which measures activity via a 3-axis algorithm. For total daytime physical activity, the measured counts of the activity tracker data minus total sleep counts were used as day-counts. Higher day-counts signify more activity. Population: Intent to treat (ITT) population: participants who received 3D regimen treatment at least once; scale down ITT (sdITT) population: excluded participants who discontinued or had missing tracker data for all study visits; modified ITT (mITT) population: excluded participants with only partial tracker data sets.
  day-counts
    sdITT Population: number analyzed (Participants) | 35
    sdITT Population | 1469569 (405329)
    mITT Population: number analyzed (Participants) | 24
    mITT Population | 1513166 (410686)
Fatigue Severity Scale (FSS) [Median (Standard Deviation); unit: score on a scale] — The FSS is a nine-item questionnaire assessing the functional impact of fatigue during the past two weeks on multiple life domains using scales from 1 (strongly disagree) to 7 (strongly agree). The fatigue score is the mean score of the 9 items, with lower scores indicating less fatigue severity. Clinically significant fatigue is usually defined as score equal or above 4. Population: Intent to treat (ITT) population: participants who received 3D regimen treatment at least once; scale down ITT (sdITT) population: excluded participants who discontinued or had missing tracker data for all study visits; modified ITT (mITT) population: excluded participants with only partial tracker data sets.
  score on a scale
    sdITT Population: number analyzed (Participants) | 37
    sdITT Population | 5.95 (0.61)
    mITT Population: number analyzed (Participants) | 24
    mITT Population | 5.94 (0.67)
Sleep Efficiency [Mean (Standard Deviation); unit: percent of time asleep] — Sleep efficiency for 2 eligible weeks (10 working days) prior to the assessment day was derived from a wrist-worn activity tracker (ActiGraph GT9X Link). Sleep efficiency was defined as the percent of time scored as sleep during the sleep period, from 0% to 100%. Population: Intent to treat (ITT) population: participants who received 3D regimen treatment at least once; scale down ITT (sdITT) population: excluded participants who discontinued or had missing tracker data for all study visits; modified ITT (mITT) population: excluded participants with only partial tracker data sets.
  percent of time asleep
    sdITT Population: number analyzed (Participants) | 35
    sdITT Population | 89.4 (4.58)
    mITT Population: number analyzed (Participants) | 24
    mITT Population | 89.8 (3.76)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Day 168 in Mean Daytime Physical Activity
Description: Mean daytime physical activity for 2 eligible weeks (10 working days) prior to the assessment day was derived from a wrist-worn activity tracker (ActiGraph GT9X Link), which measures activity via a 3-axis algorithm. For total daytime physical activity, the measured counts of the activity tracker data minus total sleep counts were used as day-counts. Higher day-counts signify more activity.
Time Frame: Baseline, Day 168
Population: ITT population: participants who received 3D regimen treatment at least once; scale down ITT (sdITT) population: excluded participants who discontinued or had missing tracker data for all study visits; modified ITT (mITT) population: excluded participants with only partial tracker data sets. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: day-counts
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 26
day-counts
  Change at Day 168: sdITT Population | -108266 (313859)
  Change at Day 168: mITT Population: number analyzed (Participants) | 24
  Change at Day 168: mITT Population | -98373 (325138)
Statistical Analysis 1: Comparison: HCV Genotype 1 Participants; sdITT (n=26): Change at Day 168 minus Baseline; Test type: Superiority; p = 0.091, one-sample t-test; mean change = -108266, 95% CI 2-sided [-235037 to 18504]
Statistical Analysis 2: Comparison: HCV Genotype 1 Participants; mITT (n=24): Change at Day 168 minus Baseline; Test type: Superiority; p = 0.152, one-sample t-test; mean change = -98373, 95% CI 2-sided [-235667 to 38921]
Statistical Analysis 3: Comparison: HCV Genotype 1 Participants; sdITT (n=26): Baseline vs. Day 168; Test type: Superiority; p = 0.091, paired t-test
Statistical Analysis 4: Comparison: HCV Genotype 1 Participants; mITT (n=24): Baseline vs. Day 168; Test type: Superiority; p = 0.152, paired t-test

2. Secondary Outcome: Change From Baseline Over Time in Mean Daytime Physical Activity
Description: as for outcome 1
Time Frame: Baseline, Days 28, 84, 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day-counts
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 34
day-counts
  Change at Day 28: sdITT Population | 26990 (211108)
  Change at Day 28: mITT Population: number analyzed (Participants) | 24
  Change at Day 28: mITT Population | 21422 (215104)
  Change at Day 84: sdITT Population: number analyzed (Participants) | 32
  Change at Day 84: sdITT Population | -6448 (198441)
  Change at Day 84: mITT Population: number analyzed (Participants) | 24
  Change at Day 84: mITT Population | -13020 (197825)
  Change at Day 168: sdITT Population: number analyzed (Participants) | 26
  Change at Day 168: sdITT Population | -108266 (313859)
  Change at Day 168: mITT Population: number analyzed (Participants) | 24
  Change at Day 168: mITT Population | -98373 (325138)
Statistical Analysis 1: Comparison: HCV Genotype 1 Participants; sdITT (n=34): Baseline vs. Day 28; Test type: Superiority; p = 0.461, paired t-test
Statistical Analysis 2: Comparison: HCV Genotype 1 Participants; mITT (n=24): Baseline vs. Day 28; Test type: Superiority; p = 0.630, paired t-test
Statistical Analysis 3: Comparison: HCV Genotype 1 Participants; sdITT (n=32): Baseline vs. Day 84; Test type: Superiority; p = 0.855, paired t-test
Statistical Analysis 4: Comparison: HCV Genotype 1 Participants; mITT (n=24): Baseline vs. Day 84; Test type: Superiority; p = 0.750, paired t-test

3. Secondary Outcome: Change From Baseline Over Time in Fatigue Severity Scale (FSS) Score
Description: The FSS is a 9-item questionnaire assessing the functional impact of fatigue during the past two weeks on multiple life domains using scales from 1 (strongly disagree) to 7 (strongly agree). The fatigue score is the mean score of the 9 items, with lower scores indicating less fatigue severity. Clinically significant fatigue is usually defined as score equal or above 4. Changes were calculated by the formula "Baseline minus Day 28, Day 84, or Day 168." Therefore the resulting negative values reflect deterioration and resulting positive values reflect improvement.
Time Frame: Baseline, Days 28, 84, 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 36
score on a scale
  Change at Day 28: sdITT Population: number analyzed (Participants) | 35
  Change at Day 28: sdITT Population | 0.69 (1.01)
  Change at Day 28: mITT Population: number analyzed (Participants) | 22
  Change at Day 28: mITT Population | 0.85 (1.06)
  Change at Day 84: sdITT Population | 1.68 (1.54)
  Change at Day 84: mITT Population: number analyzed (Participants) | 23
  Change at Day 84: mITT Population | 1.76 (1.64)
  Change at Day 168: sdITT Population | 2.60 (1.62)
  Change at Day 168: mITT Population: number analyzed (Participants) | 24
  Change at Day 168: mITT Population | 2.82 (1.52)
Statistical Analysis 1: Comparison: HCV Genotype 1 Participants; sdITT: mean change Baseline minus Day 168; Test type: Superiority; mean change = 2.60, 95% CI 2-sided [2.063 to 3.137]
Statistical Analysis 2: Comparison: HCV Genotype 1 Participants; mITT: mean change Baseline minus Day 168; Test type: Superiority; mean change = 2.82, 95% CI 2-sided [2.212 to 3.428]
Statistical Analysis 3: Comparison: HCV Genotype 1 Participants; sdITT (n=37): Baseline vs. Day 168; Test type: Superiority; p < 0.001, Paired Wilcoxon Test
Statistical Analysis 4: Comparison: HCV Genotype 1 Participants; mITT (n=24): Baseline vs. Day 168; Test type: Superiority; p < 0.001, Paired Wilcoxon Test
Statistical Analysis 5: Comparison: HCV Genotype 1 Participants; sdITT (n=35): Baseline vs. Day 28; Test type: Superiority; p < 0.001, Paired Wilcoxon Test
Statistical Analysis 6: Comparison: HCV Genotype 1 Participants; mITT (n=22): Baseline vs. Day 28; Test type: Superiority; p < 0.001, Paired Wilcoxon Test
Statistical Analysis 7: Comparison: HCV Genotype 1 Participants; sdITT (n=36): Baseline vs. Day 84; Test type: Superiority; p < 0.001, Paired Wilcoxon Test
Statistical Analysis 8: Comparison: HCV Genotype 1 Participants; mITT (n=23): Baseline vs. Day 84; Test type: Superiority; p < 0.001, Paired Wilcoxon Test

4. Secondary Outcome: Change From Baseline Over Time in Sleep Efficiency
Description: Sleep efficiency for 2 eligible weeks (10 working days) prior to the assessment day was derived from a wrist-worn activity tracker (ActiGraph GT9X Link). Sleep efficiency was defined as the percent of time scored as sleep during the sleep period, from 0% to 100%. Changes were calculated by the formula "Baseline minus Day 28, Day 84, or Day 168." Therefore the resulting negative values reflect deterioration and resulting positive values reflect improvement.
Time Frame: Baseline, Days 28, 84, 168
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of time asleep
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 34
percent of time asleep
  Change at Day 28: sdITT Population | -0.87 (2.50)
  Change at Day 28: mITT Population: number analyzed (Participants) | 24
  Change at Day 28: mITT Population | -0.44 (2.68)
  Change at Day 84: sdITT Population: number analyzed (Participants) | 32
  Change at Day 84: sdITT Population | -0.06 (2.81)
  Change at Day 84: mITT Population: number analyzed (Participants) | 24
  Change at Day 84: mITT Population | 0.01 (2.98)
  Change at Day 168: sdITT Population: number analyzed (Participants) | 26
  Change at Day 168: sdITT Population | 0.61 (3.28)
  Change at Day 168: mITT Population: number analyzed (Participants) | 24
  Change at Day 168: mITT Population | 0.74 (3.37)
Statistical Analysis 1: Comparison: HCV Genotype 1 Participants; sdITT: mean change Baseline minus Day 168; Test type: Superiority; mean change = 0.61, 95% CI 2-sided [-0.651 to 1.871]
Statistical Analysis 2: Comparison: HCV Genotype 1 Participants; mITT: mean change Baseline minus Day 168; Test type: Superiority; mean change = 0.74, 95% CI 2-sided [-0.608 to 2.088]
Statistical Analysis 3: Comparison: HCV Genotype 1 Participants; sdITT (n=37): Baseline vs. Day 168; Test type: Superiority; p = 0.381, Paired Wilcoxon Test
Statistical Analysis 4: Comparison: HCV Genotype 1 Participants; mITT (n=24): Baseline vs. Day 168; Test type: Superiority; p = 0.304, Paired Wilcoxon Test
Statistical Analysis 5: Comparison: HCV Genotype 1 Participants; sdITT (n=35): Baseline vs. Day 28; Test type: Superiority; p = 0.014, Paired Wilcoxon Test
Statistical Analysis 6: Comparison: HCV Genotype 1 Participants; mITT (n=22): Baseline vs. Day 28; Test type: Superiority; p = 0.278, Paired Wilcoxon Test
Statistical Analysis 7: Comparison: HCV Genotype 1 Participants; sdITT (n=36): Baseline vs. Day 84; Test type: Superiority; p = 0.881, Paired Wilcoxon Test
Statistical Analysis 8: Comparison: HCV Genotype 1 Participants; sdITT (n=23): Baseline vs. Day 84; Test type: Superiority; p = 0.775, Paired Wilcoxon Test

5. Secondary Outcome: Correlation Coefficients of FSS and Mean Daytime Physical Activity: sdITT Population
Description: The relationship between the parameters FSS and mean total daytime physical activity as well as for the changes of these parameters between baseline and follow-up visits was analyzed. Given a lake of normal distribution for the FSS data Spearman correlation coefficients were calculated.
Time Frame: Baseline, Days 28, 84, 168
Population: as for outcome 1
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 35
Spearman correlation coefficient
  Baseline | 0.300
  Day 28 | 0.131
  Day 84 | -0.022
  Day 168 | 0.195

6. Secondary Outcome: Correlation Coefficients of FSS and Mean Daytime Physical Activity: mITT Population
Description: as for outcome 5
Time Frame: Baseline, Days 28, 84, 168
Population: as for outcome 1
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 24
Spearman correlation coefficient
  Baseline | 0.253
  Day 28 | 0.386
  Day 84 | -0.058
  Day 168 | 0.128

7. Secondary Outcome: Correlation Coefficients of Change From Baseline Over Time in FSS and Mean Daytime Physical Activity: sdITT Population
Description: as for outcome 5
Time Frame: Baseline, Days 28, 84, 168
Population: as for outcome 1
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 34
Spearman correlation coefficient
  Baseline minus Day 28 | 0.228
  Baseline minus Day 84: number analyzed (Participants) | 32
  Baseline minus Day 84 | -0.044
  Baseline minus Day 168: number analyzed (Participants) | 26
  Baseline minus Day 168 | 0.195

8. Secondary Outcome: Correlation Coefficients of Change From Baseline Over Time in FSS and Mean Daytime Physical Activity: mITT Population
Description: as for outcome 5
Time Frame: Baseline, Days 28, 84, 168
Population: as for outcome 1
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 24
Spearman correlation coefficient
  Baseline minus Day 28 | 0.135
  Baseline minus Day 84 | -0.065
  Baseline minus Day 168 | 0.169

9. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) Post-Treatment
Description: SVR12 defined as hepatitis C virus ribonucleic acid (HCV RNA) not detectable 12 weeks after the last actual dose of paritaprevir/ritonavir/ombitasvir with dasabuvir regimen (Viekirax®/Exviera®, 3D regimen).
Time Frame: Day 168 (or 12 weeks after the last dose of study drug)
Population: ITT population: participants who received 3D regimen treatment at least once; scale down ITT (sdITT) population: excluded participants who discontinued or had missing tracker data for all study visits; modified ITT (mITT) population: excluded participants with only partial tracker data sets.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCV Genotype 1 Participants
Number analyzed (Participants) | 41
percentage of participants
  ITT Population | 97.6 [95.2 to 100]
  sdITT Population: number analyzed (Participants) | 37
  sdITT Population | 97.3 [92.3 to 100]
  mITT Population: number analyzed (Participants) | 24
  mITT Population | 95.8 [88.3 to 100]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Day 168
Arm/Group | HCV Genotype 1 Participants
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 9/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCV Genotype 1 Participants (N=41)
Nausea (Gastrointestinal disorders) | 6 (6)
Dizziness (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03002818/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03002818/SAP_001.pdf